CLINICAL TRIAL: NCT03741348
Title: Erector Spinae Plane Block For Postoperative Analgesia in Patients Undergoing Total Abdominal Hysterectomy: A Randomized Controlled Study
Brief Title: Erector Spinae Plane Block For Postoperative Analgesia in Patients Undergoing Total Abdominal Hysterectomy
Acronym: Erector Spinae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mohamed hamed, lecturer of anesthesia, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R124
Record Dates: First submitted 2018-11-11; First posted 2018-11-14 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Pain
Keywords: Erector Spinae Plane Block; Postoperative Analgesia; Total Abdominal Hysterectomy; fentanyl consumption
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ES (Active Comparator): Erector Spinae Plane Block
  Interventions: Procedure: Erector Spinae Plane Block
- control (Placebo Comparator): the control group will not receive block
  Interventions: Procedure: control

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — In (ES) group After skin sterilization, ESPB was performed in sitting position at the level of T9 linear ultrasound (US) transducer (Phillips-Saronno Italy) was placed vertically 3cm lateral to midline to visualize the muscles of the back, transverse process and simmering pleura in between the two transverse processes. After local infiltration of needle insertion site with 2-3ml of 2% lidocaine, a 22-gauge Short bevel needle (Spinocan, B.Braun Melsungen AG, Germany) was inserted in cranial-caudal direction towards transverse process (TP) in-plane to the US transducer until needle touched the TP crossing all the muscles. Then, up to 20 ml of bupivacaine 0.5% was injected. The procedure was repeated following the same steps on the other side of back.
  Arms: ES
Procedure: control — in control group, Erector Spinae Plane Block will not be done
  Arms: control

SUMMARY:
The aim of this study was to assess the efficacy of bilateral ESPB on postoperative analgesia in patients undergoing total abdominal hysterectomy under general anesthesia.

DETAILED DESCRIPTION:
60 patients Scheduled for elective total abdominal hysterectomy, after obtaining a written informed consent for anesthesia from each patient before enrolment in the study after explaining to them the nature of study.

Inclusion criteria included female patients aged 40 - 70 years, Weighted 50 - 90 Kg and with American society of anesthesiologists physical status (ASA) class Ι to ΙΙΙ Scheduled for elective total abdominal hysterectomy under general anesthesia. Exclusion criteria included Local infection at the site of puncture, Patients having history of hematological disorders, including coagulation abnormality, Patients with severe hepatic impairment, Patients with chronic pain and Patient had a known allergy to study drugs.

Patients were randomized into two equal groups. An online randomization program was used to generate random number list. Patient randomization numbers were concealed in opaque envelops which were opened by the study investigator.

Members of the study group involved in obtaining functional data were blinded to randomization for the period of data acquisition and analysis. Patients were randomly allocated into two groups:

Erector spinae plane block Group (ES): ultrasound guided erector spinae plane block at T9 vertebrae level with 20 ml of bupivacaine 0. 5%. Control Group (c): did not receive block.

One day before surgery all patients were interviewed to explain visual analogue scale (VAS), learned how to use patient controlled analgesia (PCA) pump and routine investigations were fulfilled.

In both groups Patients were monitored with ECG, non-invasive blood pressure monitoring and pulse oximetry. IV access was established and IV midazolam 0.01-0.02 mg.kg-1 was given.

In (ES) group After skin sterilization, ESPB was performed in sitting position at the level of T9 linear ultrasound (US) transducer (Phillips-Saronno Italy) was placed vertically 3cm lateral to midline to visualize the muscles of the back: the trapezius muscle above, the rhomboid major muscle in the middle and the erector-spinae muscle on the bottom, transverse process and simmering pleura in between the two transverse processes. After local infiltration of needle insertion site with 2-3ml of 2% lidocaine, a 22-gauge Short bevel needle (Spinocan, B.Braun Melsungen AG, Germany) was inserted in cranial-caudal direction towards transverse process (TP) in-plane to the US transducer until needle touched the TP crossing all the muscles. Correct needle placement was confirmed by Visualizing the needle in plane along its entire length, when it contacted the transverse process, 1 ml of anesthetic solution was injected. Hydrodissection of the interfascial plane between the erector spinae muscle and the transverse process was confirmed by visualizing the local anesthetic spreading in a linear pattern between the muscle and the bony acoustic shadows of the transverse process, ensuring correct localization. Then, up to 20 ml of bupivacaine 0.5% was injected. The procedure was repeated following the same steps on the other side of back. Control Group (c): the same pervious technique as in ES group but patient did not receive block.

Block success was tested by reduced cold sensation at planned surgical incision 5 minutes after block completion.

General anesthesia was induced with fentanyl 2 mcg.kg-1, propofol 2 mg.kg-1 followed by atracium 0.5 mg.kg-1 and after intubation Anesthesia was maintained with isoflurane (1 MAC) and atracium 0.1mg.kg-1 as a maintenance dose every 30 minutes till the end of the procedure; After emerging from anesthesia, the patients were transferred to the post aesthesia care unit (PACU) for a 2 hours observation period. The patients were discharged from the PACU after fulfilling the discharge criteria based on Aldrete score. Postoperative analgesia was provided in both groups immediately after surgery by PCA fentanyl pump then regular oral acetaminophen 1 g four times a day.

The criteria to stop fentanyl titration protocol were satisfactory pain control, Patient became sedated (Ramsay sedation scale >2), Respiratory rate < 12 / min, Oxygen saturation < 95% or development of serious adverse effects (allergy, severe vomiting, hypotension).

Visual analogue pain score (VAS) for pain (ranging from 0 to 10, where 0 no pain and 10 maximum pain) was measured postoperatively at 30 min and 2, 4, 6, 12, and 24 hour postoperative.

Any side effects were recorded as nausea or vomiting, pneumothorax, or any other complications. Also Duration of hospital stays, from the first day postoperative until discharge.

The primary outcome of this study was Total fentanyl consumption in the first 24 hours And The secondary outcome was VAS for pain (ranging from 0 to 10, where 0 no pain and 10 maximum pain) was evaluated postoperatively at 30 min and 2, 4, 6, 12, and 24 hour postoperative, Duration of hospital stays and any complications.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* Aged 40 - 70 years,
* Weighted 50 - 90 Kg
* American society of Anesthesiologists physical status (ASA) class Ι to ΙΙΙ
* Scheduled for elective total abdominal hysterectomy under general anesthesia

Exclusion Criteria:

* Local infection at the site of puncture
* Patients having a history of hematological disorders, including coagulation abnormality
* Patients with severe hepatic impairment
* Patients with chronic pain
* A patient had a known allergy to study drugs.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Fentanyl consumption | first 24 hours postoperative
  in microgram

SECONDARY OUTCOMES:
Visual analog score | 30 minutes postoperative
  ranging from 0 to 10, where 0 no pain and 10 maximum pain
Visual analog score | 2 hours postoperative
  ranging from 0 to 10, where 0 no pain and 10 maximum pain
Visual analog score | 4 hours postoperative
  ranging from 0 to 10, where 0 no pain and 10 maximum pain
Visual analog score | 6 hours postoperative
  ranging from 0 to 10, where 0 no pain and 10 maximum pain
Visual analog score | 12 hours postoperative
  ranging from 0 to 10, where 0 no pain and 10 maximum pain
Visual analog score | 24 hours postoperative
  ranging from 0 to 10, where 0 no pain and 10 maximum pain

OTHER OUTCOMES:
Age | 4 hours before operation once recruited
  in years
Weight | 4 hours before operation once recruited
  in Kilogram
Duration of surgery | 4 minutes after end of operation
  in minutes

CONTACTS AND LOCATIONS:
Overall Officials: mohamed a hamed, MD, Principal Investigator — Fayoum University
Locations (1):
- Mohamed, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azari L, Santoso JT, Osborne SE. Optimal pain management in total abdominal hysterectomy. Obstet Gynecol Surv. 2013 Mar;68(3):215-27. doi: 10.1097/OGX.0b013e31827f5119. PMID 23945838
- [Background] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158
- [Background] Ueshima H, Otake H. Similarities Between the Retrolaminar and Erector Spinae Plane Blocks. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):123-124. doi: 10.1097/AAP.0000000000000526. No abstract available. PMID 27997492